CLINICAL TRIAL: NCT05514821
Title: Effects of Dietary Nitrate on Blood Pressure: Exploring the Repeatability and Inter-individual Variation in Responses
Brief Title: Inter-individual Variation in the Blood Pressure Lowering Effects of Dietary Nitrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: University of the West of Scotland (Other); University of Nottingham (Other); Aspire Academy (Other Government); Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NU013253
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Blood Pressure
Keywords: Hypertension; Personalized nutrition; Nitric oxide; Beetroot juice
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Replicated cross-over trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplements will be administered double blind (participant and researcher blind) in identical bottles. They will be identical in smell, taste, texture and colour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental condition 1 (Experimental): Acute supplementation with 140 ml Beet It Sport Shots, James White Ltd (~400mg dietary nitrate)
  Interventions: Dietary Supplement: Beet It Sport Shot
- Experimental condition 2 (Experimental): Acute supplementation with 140 ml Beet It Sport Shots, James White Ltd (~400mg dietary nitrate)
  Interventions: Dietary Supplement: Beet It Sport Shot
- Control condition 1 (Placebo Comparator): Acute supplementation with 140 ml nitrate-depleted Beet It Sport Shots, James White Ltd (~0mg dietary nitrate)
  Interventions: Dietary Supplement: Beet It Sport Shot Placebo
- Control condition 2 (Placebo Comparator): Acute supplementation with 140 ml nitrate-depleted Beet It Sport Shots, James White Ltd (~0mg dietary nitrate)
  Interventions: Dietary Supplement: Beet It Sport Shot Placebo

INTERVENTIONS:
Dietary Supplement: Beet It Sport Shot — Acute supplementation with 140 ml Beet It Sport Shots, James White Ltd, containing ~400mg dietary nitrate
  Arms: Experimental condition 1; Experimental condition 2
Dietary Supplement: Beet It Sport Shot Placebo — Acute supplementation with 140 ml Beet It Sport Shots Placebo, James White Ltd, in which the nitrate has been removed via an ion exchange resin, containing ~ 0 mg dietary nitrate
  Arms: Control condition 1; Control condition 2

SUMMARY:
Dietary nitrate supplementation, often in the form of beetroot juice, has been shown to lower blood pressure and could play a role in preventing or treating hypertension. However, it is currently unclear: a) how reproducible this response is within the same individual on different occasions, and b) whether there are genuine individual differences in the blood pressure lowering effects of dietary nitrate. This study will use a novel replicated cross-over design (2 x nitrate conditions, 2 x placebo conditions) to examine the reproducibility and inter-individual variability in the blood pressure lowering effects of dietary nitrate supplementation.

DETAILED DESCRIPTION:
The investigators will undertake a replicated cross-over randomised controlled trial (i.e., a study involving 2 x identical experimental conditions and 2 x identical control conditions), to explore the reproducibility of the blood pressure lowering effects of nitrate-rich beetroot juice, and to identify if there are genuine individual differences in the blood pressure-lowering effects of this supplement. Participants will be recruited via posters, email and social media, and interested individuals will be invited to attend the laboratory on 5 occasions.

Visit 1: Potential participants will be invited to attend a screening session at Newcastle University to identify if they are eligible to participate. They will have an opportunity to discuss the study with a researcher and will provide written consent. They will then complete a screening questionnaire and provide a measure of their height, weight and blood pressure. Eligible participants will be invited to attend 4 experimental trials (2 x nitrate-rich beetroot juice conditions, 2 x placebo conditions) over 2-3 weeks with a minimum of 3 days wash-out between visits. If individuals are ineligible to participate this will be explained to them and they will be thanked for their time.

Visits 2-5: On the day before the first trial, participants will be asked to record what they eat and then replicate this as closely as possible for all future visits. In the morning of each trial, participants will be asked to arrive at the laboratory between 7-9 am having fasted since 10 pm the night before. The participants will be required to rest for 10 minutes, after which a measure of their blood pressure will be obtained. Participants will then be provided with breakfast (a bowl of porridge) and 140 ml concentrated nitrate-rich (~12.5 mmol nitrate) or nitrate-depleted beetroot juice (~0 mmol nitrate). Participants will then be asked to sit in the laboratory for 2.5 hours, during which time they can read quietly or use a computer. The investigators will then obtain a further measure of their blood pressure and collect a blood sample from a vein in their arm via venepuncture, to measure markers of nitric oxide, a signalling molecule in the body which is thought to mediate the blood pressure lowering effects of nitrate-rich beetroot juice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Aged 18 - 45 years

Exclusion Criteria:

* Aged less than 18 or more than 45 years old
* Female
* Currently taking any medication or antibiotics
* Attending general practitioner for a health problem or on a hospital waiting list
* Currently taking part in another research study which could conflict with the requirements for this investigation
* Regularly use antibacterial mouthwash and unwilling to stop using this throughout the study period
* Current smoker
* History of kidney, liver or cardiovascular disease
* Have diabetes
* Have a gastrointestinal disorder
* Recent history (past 1 year) of cancer
* Use of other dietary supplements e.g., pre and probiotics
* Currently dieting
* Have a known allergy to any components within the dietary supplement

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Blood pressure of the brachial artery | Immediately prior to supplementation and for 2.5 hours after supplementation
  Blood pressure of the brachial artery

SECONDARY OUTCOMES:
Plasma nitrite concentrations | 2.5 hours after supplementation
  Plasma nitrite concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Shannon, PhD, Principal Investigator — Newcastle University
Locations (1):
- Human Nutrition & Exercise Research Centre, Newcastle upon Tyne, Northumberland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to a repository following publication of the study results
Time Frame: Within 6 months of publication of the study findings

REFERENCES:
- [Derived] Hayes E, Alhulaefi S, Siervo M, Whyte E, Kimble R, Matu J, Griffiths A, Sim M, Burleigh M, Easton C, Lolli L, Atkinson G, Mathers JC, Shannon OM. Inter-individual differences in the blood pressure lowering effects of dietary nitrate: a randomised double-blind placebo-controlled replicate crossover trial. Eur J Nutr. 2025 Feb 24;64(2):101. doi: 10.1007/s00394-025-03616-x. PMID 39992469